CLINICAL TRIAL: NCT07119268
Title: SPARK-Healthy Sleep: A Digital Health Intervention to Promote Behavioral, Emotional, and Cognitive Changes
Brief Title: SPARK Healthy Sleep
Acronym: SPARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Principal Investigator, Kyle S. Minor, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPARK Healthy Sleep
Record Dates: First submitted 2025-07-31; First posted 2025-08-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia and Related Disorders; Sleep Disturbance
Keywords: College Students; Sleep Disturbances; Psychosis-Spectrum Disorders
MeSH Terms: conditions — Schizophrenia; Parasomnias

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 into two groups that run simultaneously (in parallel)
  Experimental Group: Receives SPARK-Healthy Sleep intervention immediately at baseline Control Group: Wait-list control that receives the intervention after a 3-week delay (after the study's primary endpoint)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Experimental Group (Experimental): Receives SPARK-Healthy Sleep intervention immediately at baseline
  Interventions: Device: SPARK Healthy Sleep
- Control Group (No Intervention): Wait-list control that receives the intervention after a 3-week delay (after the study's primary endpoint)

INTERVENTIONS:
Device: SPARK Healthy Sleep — SPARK-Healthy Sleep is a single-session digital intervention delivered via smartphone that combines stigma reduction with evidence-based sleep improvement strategies.
  Arms: Experimental Group

SUMMARY:
SPARK-Healthy Sleep is a digital mental health intervention designed to help college students who may be at risk for psychosis and experience sleep problems. About 1 in 4 college students report psychotic-like experiences (such as hearing voices or feeling paranoid), and these students often have poor sleep quality, which can worsen their mental health symptoms.

This study tests whether a single-session digital intervention can improve sleep and reduce mental health stigma in at-risk college students. The intervention is delivered through a smartphone app and takes about 30 minutes to complete. It includes educational content about mental health being on a continuum (not just "normal" vs "abnormal"), strategies to reduce stigma around seeking help, and evidence-based sleep improvement techniques based on cognitive behavioral therapy for insomnia.

The study will recruit 115 college students from Indiana University-Indianapolis who score high on measures of psychotic-like experiences and poor sleep quality. Half will receive the intervention immediately (experimental group), while the other half will wait three weeks before receiving it (control group). All participants will complete questionnaires about sleep, mental health symptoms, social functioning, and stigma at the beginning of the study and after two weeks.

The main goals are to determine if the intervention is feasible and acceptable to students, and whether it shows preliminary effectiveness in improving sleep quality, reducing stigma, and improving overall mental health outcomes. A subset of participants will also complete interviews about their experience using the intervention.

This research addresses important barriers to mental health care for college students, including stigma and limited access to services. If successful, this digital approach could provide a scalable way to help at-risk students improve their mental health and potentially prevent more serious problems from developing.

DETAILED DESCRIPTION:
Study Overview SPARK-Healthy Sleep is a randomized controlled pilot study testing a single-session digital mental health intervention for college students at risk for psychosis who experience sleep difficulties. The study evaluates feasibility, acceptability, and preliminary effectiveness of a smartphone-delivered intervention combining stigma reduction and cognitive behavioral therapy for insomnia (CBT-I) principles.

Study Design This is a pragmatic randomized controlled trial with a wait-list control design. Participants are randomized 1:1 to immediate intervention or 3-week delayed intervention, stratified by race, gender, and age. The study is unblinded given the nature of the digital intervention.

Participants and Recruitment Target enrollment: 115 college students from Indiana University-Indianapolis (aiming for 100 completers). Recruitment occurs through the SONA research participation system and mass emails to the student body.

Inclusion Criteria: Age ≥18 years, Current college enrollment, English fluency, Prodromal Questionnaire-Brief endorsement score ≥7, Pittsburgh Sleep Quality Index score >5, Pass validity screening questions

Exclusion Criteria: Previous psychotic disorder diagnosis, Unable to provide informed consent

Intervention Description

SPARK-Healthy Sleep is delivered via Qualtrics platform in approximately 30 minutes. The intervention consists of five modules:

Introduction: Welcome, safety information, single-session concept introduction Stigma Resistance: Mental health continuum education, stress-vulnerability model, interactive exercises Sleep Regulation: CBT-I principles, sleep hygiene education, cognitive restructuring, behavioral strategies Planning: Personalized sleep plan development, goal-setting exercises Recap: Summary, resource provision, follow-up instructions

The intervention incorporates videos, interactive text responses, and personalized feedback based on participant inputs.

Assessment Schedule

Screening Assessment:

Online consent process Demographics questionnaire Schizotypal Personality Questionnaire-Brief Updated Prodromal Questionnaire-Brief Pittsburgh Sleep Quality Index Additional measures: Academic satisfaction, life satisfaction, loneliness, digital mental health interest

Baseline Assessment (Week 0):

Comprehensive battery including sleep quality, stigma measures, affect, paranoid ideation, social functioning, depression, emotion regulation, and cognitive testing Intervention installation and orientation for experimental group

Follow-up Assessment (Week 2):

Repeat of baseline measures System usability and intervention acceptability measures Intervention access provided to control group

Qualitative Interviews:

Semi-structured interviews with 10 participants selected across engagement levels Audio recorded with permission Focus on user experience, barriers, and improvement suggestions

Primary Outcomes Feasibility: Intervention completion rates (target ≥80%), system usability scores Acceptability: Intervention appropriateness ratings, prompt completion rates Usage data: Time spent, modules completed, interaction frequency

Secondary Outcomes Sleep quality (Pittsburgh Sleep Quality Index) Mental health stigma (Internalized Stigma Mental Health Inventory) Paranoid ideation (Community Assessment of Psychic Experiences) Negative affect (Positive and Negative Affect Schedule) Functional outcomes: Social functioning, depression, emotion regulation, executive functioning

Statistical Analysis Plan Sample Size: Power analysis indicates n=50 per arm provides adequate power (0.80) to detect medium effects (α=0.05).

Primary Analysis: Descriptive statistics for feasibility and acceptability outcomes. Target thresholds: ≥80% completion rates and high usability/appropriateness ratings.

Secondary Analysis: 2x2 mixed-effects ANOVA examining intervention effects over time (baseline, follow-up) and between conditions (immediate vs. delayed intervention). Within-group effect sizes calculated to quantify intervention impact. Bonferroni corrections applied for multiple comparisons.

Missing Data: Multiple imputation for missing at random data. Intent-to-treat analysis with sensitivity analyses for different missingness patterns.

Qualitative Analysis: Thematic content analysis of interview transcripts to identify implementation barriers and improvement recommendations.

Data Management and Quality Assurance Data Collection: All data collected via password-protected Qualtrics surveys stored on secure IU research servers.

Quality Control:

Range checks in Qualtrics Double entry for critical variables Regular data backup verification Monthly data quality review by PI

Safety Monitoring:

Automated flags for concerning responses on depression and psychosis measures 24-hour PI notification protocol Established referral pathways to campus counseling and first-episode psychosis services Resource information provided to all participants

Data Storage: De-identified data stored indefinitely on encrypted servers. Separate master list links participant IDs to identifying information, accessible only to PI and study team.

This pilot study will provide essential feasibility data and preliminary effect size estimates for future larger-scale randomized controlled trials examining longer-term outcomes and broader implementation across college campuses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Current college enrollment
* English fluency
* Prodromal Questionnaire-Brief endorsement score ≥7
* Pittsburgh Sleep Quality Index score >5
* Pass validity screening questions

Exclusion Criteria:

* Previous psychotic disorder diagnosis
* Unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Intervention Completion Rates | 2 weeks
System Usability Scores | 2 weeks
Intervention Appropriateness Ratings | 2 weeks
Prompt Completion Rates | 2 weeks
Time Spent on Modules | 2 weeks
  Total amount of time spent on modules over two weeks
Interaction Frequency | 2 weeks
  Number of times engaging with intervention

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 2 weeks
  Sleep quality
Internalized Stigma Mental Health Inventory | 2 weeks
  Stigma
The Community Assessment of Psychic Experiences (CAPE) | 2 weeks
  Paranoia questionnaire (42 items)
Positive and Negative Affect Schedule | 2 weeks
  Affect
Social Functioning Scale | 2 weeks
  Social functioning
Beck Depression Inventory | 2 weeks
  Depression

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided